CLINICAL TRIAL: NCT02216058
Title: A Prospective, Multicenter Trial of NOYA Sirolimus-Eluting Stent With Biodegradable Coating in Patients With Coronary Artery Disease
Brief Title: Safety and Efficacy Study of NOYA Sirolimus-Eluting Stent to Treat Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medfavour (Beijing) Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WR-CT-001
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NOYA (Experimental): NOYA CoCr Biodegradable Coating Sirolimus-Eluting Stent System
  Interventions: Device: NOYA CoCr Biodegradable Coating Sirolimus-Eluting Stent System

INTERVENTIONS:
Device: NOYA CoCr Biodegradable Coating Sirolimus-Eluting Stent System

SUMMARY:
A prospective, multicenter study is preformed to evaluate the safety and efficacy of NOYA CoCr biodegradable coating sirolimus-eluting stents in treating coronary artery lesions.

DETAILED DESCRIPTION:
A prospective, multicenter study is preformed to evaluate the safety and efficacy of NOYA CoCr biodegradable coating sirolimus-eluting stents in treating coronary artery lesions. Appropriate patients judged by inclusion and exclusion standards will be preformed stent implantation, and after that all patients will be clinically followed up at 30, 180, 365 days,2 years,3 years,4 years and 5 years. Target Lesion Failure (TLF) found in following-up period as key indicators to evaluate the safety of stents. The arrangement, conclusion and statistical analysis of trial data including clinography and angiography will be fulfilled by independent Data Management Center(DMC) and radiography core laboratory.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥18 of age; male or non-pregnant female.
* Diagnosis of coronary artery disease.
* At least one target lesion with a diameter stenosis ≥70% (visual estimate)
* Acceptable candidate for CABG;
* The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written Notice of Informed Consent, appropriate Ethics Committee(EC); and the patient is willing to comply with specified follow-up evaluations.

Exclusion Criteria:

* Patient has congenital heart disease, severe valve dysfunction, bridge vascular disease, severe heart failure (NYHA ≥ Ⅲ level), or left ventricular ejection fraction ≤ 30%.
* Patient has undergone previous stenting anywhere within the previous 1 year. Patient has a preoperative renal dysfunction: serum creatinine> 2.0mg/dl (176.82umol / L).
* Patient has a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated or in which patient will not be able to comply with dual antiplatelet therapy for at least 1 year;
* Patient has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, clopidogrel/ticlopidine, Prasugrel, stainless steel alloy, cobalt chromium, rapamycin, styrene-butylene-styrene or poly-lactic acid (PLA) polymer, and/or contrast sensitivity that cannot be adequately premedicated;
* Patient is allergic to contrast agent Sirolimus.
* Patient has a limited life expectancy is less than 12 months.
* Currently participating in another investigational drug or device study or patient in inclusion in another investigational drug or device study during follow-up.
* Patient has poor compliance with the judgment of the investigator and can not complete the study as required.
* Patient who had heart transplant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
TLF(Target Lesion Failure) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Dr., Principal Investigator — Chines PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China